CLINICAL TRIAL: NCT01834157
Title: The "DeSScipher" Project - to Decipher the Best Treatment for Systemic Sclerosis - Observational Trial 2: Improvement of Hand Dysfunction by Arthritis in Systemic Sclerosis
Brief Title: Improvement of Hand Dysfunction by Arthritis in Systemic Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prof. Laszlo Czirjak (Other)
Collaborators: European Union (Other); University of Giessen (Other); University of Zurich (Other); University of Paris 5 - Rene Descartes (Other); University of Florence (Other); University of Campania Luigi Vanvitelli (Other); University of Basel (Other); University College, London (Other); Charite University, Berlin, Germany (Other); University of Leeds (Other); Schoen Klinik Hamburg Eilbek (Other)
Responsible Party: Sponsor-Investigator, Prof. Laszlo Czirjak, Prof. Laszlo Czirjak, University of Pecs
Organization: University of Pecs (Other)
Other Study IDs: HEALTH-F5-2012-305495-OT2
Record Dates: First submitted 2013-04-09; First posted 2013-04-17 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Systemic Sclerosis; Arthritis
MeSH Terms: conditions — Scleroderma, Systemic; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- methotrexate: methotrexate with or without low-dose corticosteroids
- other DMARDs: other DMARDs (leflunomide, azathioprine, mycophenolate mofetil) with or without low-dose corticosteroids
- low-dose corticosteroids: low-dose corticosteroids without DMARDs
- No DMARD or corticosteroids: No DMARD or corticosteroid treatment
- CPH/CSA - Exploratory cohort: cyclophosphamide or cyclosporine-A with or without other DMARDs or low-dose corticosteroids
- Biologics - Exploratory cohort: Biologic therapy with or without other DMARDs or low-dose corticosteroids
- Combinations - Exploratory cohort: Combination of two or more DMARDs with or without low-dose corticosteroids

SUMMARY:
Systemic sclerosis (SSc) is an orphan, multiorgan disease affecting the connective tissue of the skin and several internal organs. Beside skin involvement, digital ulcers, tendinitis, calcinosis and flexion contractures, the presence of hand arthritis is a major contributor to impairment of hand function in systemic sclerosis. Several immunomodulatory drugs used in other rheumatic diseases (including methotrexate, leflunomide, azathioprine, mycophenolate mofetil and low-dose corticosteroids) can potentially improve arthritis and consequently hand function in systemic sclerosis. For the assessment of arthritis, the CDAI (clinical disease activity index) is validated in rheumatoid arthritis, and may be useful for SSc-related arthritis, too.

This observational trial is part of the collaborative project "DeSScipher", one out of five observational trials to decipher the optimal management of systemic sclerosis. Aim of this observational trial is to:

* investigate the efficacy and safety of different treatments on hand dysfunction in systemic sclerosis patients with hand arthritis and
* to validate the CDAI for arthritis in systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile and adult Systemic sclerosis patients, with diagnosis according to the ACR/EULAR adult SSc criteria and PRES/ACR/EULAR juvenile SSc criteria respectively
* Clinical signs of arthritis (defined as ≥2 tender and swollen joints)

Exclusion Criteria:

* Presence of significant, long standing articular pain due to other cause than autoimmune disease
* Presence of hand disability caused by other, than autoimmune disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is adult and juvenile systemic sclerosis patients from the EUSTAR cohort (MEDSonline database) and the jSScWG cohort.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Improvement of HAQ-DI (CHAQ-DI in jSSc) by at least -0.21 in one year | 12 months
  Improvement from baseline in Health Assessment Questionnaire - Disability Index (Child Health Assessment Questionnaire - Disability Index in juvenile systemic sclerosis) by at least -0,21(moderate improvement) in one year

SECONDARY OUTCOMES:
Improvement of the CHFS in one year | 12 months
  Improvement of the Cochin Hand Function Scale in one year
Improvement of the CDAI in one year | 12 months
  Improvement of the Clinical Disease Activity Index in one year
Improvement of the SDAI in one year | 12 months
  Improvement of the Simplified Disease Activity Index in one year
Improvement of the DAS28(We) in one year | 12 months
  Improvement of the Disease Activity Score 28 (using 4 variables, including erythrocyte sedimentation rate) in one year
Improvement of the DAS28(CRP) in one year | 12 months
  Improvement of the Disease Activity Score 28 (using 4 variables, including C-reactive protein) in one year

OTHER OUTCOMES:
Validation of the CDAI in systemic sclerosis | 12 months
  Exploratory endpoint: Validation of the Clinical Disease Activity Index in systemic sclerosis
Validation of the SDAI in systemic sclerosis | 12 months
  Exploratory endpoint: Validation of the Simplified Disease Activity Index in systemic sclerosis
Validation of the DAS28(ESR) in systemic sclerosis | 12 months
  Exploratory endpoint: Validation of the Disease Activity Score 28 (using 4 variables, including erythrocyte sedimentation rate) in systemic sclerosis
Validation of the DAS28(CRP) in systemic sclerosis | 12 months
  Exploratory endpoint: Validation of the Disease Activity Score 28 (using 4 variables, including C-reactive protein) in systemic sclerosis
Evaluation of the incidence and potential predictors of deterioration of hand dysfunction and progression of arthritis in systemic sclerosis | 24 months
  Evaluation of the incidence and potential predictors of deterioration of hand dysfunction and progression of arthritis in systemic sclerosis
Incidence of drug-related adverse events | 24 months
  Evaluation of the incidence of drug-related adverse events
Incidence of withdrawal from treatment due to drug-related adverse events | 24 months
  Evaluation of the incidence of withdrawal from treatment due to drug-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Müller-Ladner, Prof., Study Chair — Justus-Liebig-University Gießen, Kerckhoff Clinic, Departement of Rheumatology and Clinical Immunology; Laszlo Czirjak, Prof, Principal Investigator — PECSI TUDOMANYEGYETEM - UNIVERSITY OF PECS
Locations (33):
- University of Ghent, Department of Rheumatology, Ghent, Belgium
- Dubrava University Hospital, Zagreb, Croatia
- Assiut and Sohage University Hospital Rheumatology Department Assiut University Hospital, Asyut, Egypt
- France (2):
  - Department of Internal Medicine Hôpital Claude Huriez, Lille
  - Université Paris Descartes, Hôpital Cochin, Service de Rhumatologie A & INSERM 1016, Paris
- Germany (8):
  - Justus-Liebig-University Gießen, Kerckhoff Clinic, Departement of Rheumatology and Clinical Immunology, Bad Nauheim
  - Charité Universitätsmedizin Berlin, Charité Centrum 12 für Innere Medizin und Dermatologie, Medizinische Klinik mit Schwerpunkt Rheumatologie und Klinische Immunologie, Berlin
  - Universitätshautklinik Köln, Cologne
  - Universitätsklinikum Erlangen, Erlangen
  - Endokrinologikum Frankfurt, Frankfurt
  - Centre for Pediatric Rheumatology, Klinikum Eilbek, Hamburg
  - Medizinische Universitätsklinik Abt. II, Tübingen
  - Krankenhaus St. Josef, Wuppertal
- Pecsi Tudomanyegyetem - University of Pecs, Pécs, Hungary
- Italy (6):
  - Istituto di Clinica Medica Generale, Ematologia ed Immunologia Clinica, Università Politecnica delle Marche, Polo Didattico, University of Ancona, Ancona
  - University of Florence, Denothe Centre, Division of Rheumatology AOUC, Department of Biomedicine, Florence
  - Department of Rheumatology, University of Cagliari-Policlinico Universitario, Monserrato
  - Policlinico, Via Pansini, Napoli-Italia
  - University of Padova, Padua
  - Divisione di Reumatologia, Università di Roma La Sapienza, Dipartimento di Clinica e Terapia medica applicata, Policlinico Umberto I, Roma
- Romania (3):
  - Department of Internal Medicine and Rheumatology Clinic, Ion Cantacuzino Clinical Hospital, Bucharest
  - Reumatologie, University of Medicine & Pharmacy,"Iuliu Hatieganu" Cluj, Cluj-Napoca
  - GR.T.Popa Center for Biomedical Research, European Center for Translational Research, "GR.T.Popa" University of Medicine and Pharmacy, Rehabilitation Hospital, Iași
- Russia (2):
  - Clinic of Nephrology, Internal and Occupational Diseases, Moscow
  - Institute of Rheumatology, Russian Academy of Medical Science, Moscow
- Institute of Rheumatology Belgrade, Belgrade, Serbia
- Hospital Universitario Madrid Norte Sanchinarro, Madrid, Spain
- Switzerland (2):
  - Felix-Platter Spital, Basel
  - University of Zurich, Department of Rheumatology, Zurich
- University of Marmara, Department of Rheumatology, Istanbul, Turkey (Türkiye)
- United Kingdom (3):
  - The Universitiy of Leeds, Division of Rheumatic and Musculoskeletal Disease, St James's University Hospital, Leeds
  - Royal Free Hospital, University College London, London
  - University of Manchester, Rheumatic Diseases Centre, Clinical Sciences, Manchester,Salford